CLINICAL TRIAL: NCT01271413
Title: Effects of Cognitive Training in Methadone Maintenance Patients
Brief Title: Cognitive Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Miriam Mintzer, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00042772; 1R21DA029708 (NIH)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive cognitively stimulating activities (Experimental)
  Interventions: Behavioral: Computerized cognitively stimulating activities
- Non-adaptive cognitively stimulating activities (Active Comparator)
  Interventions: Behavioral: Computerized cognitively stimulating activities

INTERVENTIONS:
Behavioral: Computerized cognitively stimulating activities — The study will compare the effects of different methods of computerized mental stimulation. The intervention involves 25 sessions involving computerized cognitive tasks.

SUMMARY:
This research is being done to learn if computer tasks that challenge the brain (cognitively stimulating tasks) can improve memory and other types of thinking. The study will compare the effects of different versions of the computer tasks. It also will compare the task performance of different groups of people.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* in methadone maintenance or healthy volunteers
* healthy

Exclusion Criteria:

* Axis I disorder (except substance abuse and dependence in methadone maintenance patients)
* severe cognitive impairment
* serious untreated medical condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2010-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Z Mintzer, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- BPRU, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Rass O, Schacht RL, Buckheit K, Johnson MW, Strain EC, Mintzer MZ. A randomized controlled trial of the effects of working memory training in methadone maintenance patients. Drug Alcohol Depend. 2015 Nov 1;156:38-46. doi: 10.1016/j.drugalcdep.2015.08.012. Epub 2015 Aug 24. PMID 26404954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adaptive Cognitively Stimulating Activities | Non-adaptive Cognitively Stimulating Activities
Started | 37 | 36
Completed | 28 | 28
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Cognitively Stimulating Activities; Cognitively Stimulating Activities: Other: Computerized cognitively stimulating activities: The study will compare the effects of different methods of computerized mental stimulation. The intervention involves 25 sessions involving computerized cognitive tasks.
- Total: Total of all reporting groups
Arm/Group | Cognitively Stimulating Activities | Cognitively Stimulating Activities: Other | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (8.8) | 43.5 (7.1) | 43.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Working Memory
Description: Change in maximum number of digits correctly recalled in Digit Span Backwards task, from baseline to 7 weeks
Time Frame: baseline, 7 weeks
Measure: Mean (Standard Deviation); unit: digits recalled
Arm/Group | Adaptive Cognitively Stimulating Activities | Non-adaptive Cognitively Stimulating Activities
Number analyzed (Participants) | 28 | 28
digits recalled | 0.86 (1.21) | 0.04 (0.92)

2. Secondary Outcome: Episodic Memory
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Trail-making
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

4. Secondary Outcome: go/No-go
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Addiction Severity Index
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Delay Discounting
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Digit Symbol Substitution Test
Time Frame: baseline, 7 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cognitively Stimulating Activities | Cognitively Stimulating Activities: Other
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes